CLINICAL TRIAL: NCT00448513
Title: Effects of Tea Catechin Extracts on the Frequency Changes of Micronuclei in Peripheral Lymphocytes in Late Middle Aged Healthy Volunteers
Brief Title: Effects of Tea Catechin Extracts on Oxidative Damage
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Shizuoka (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: CT2006005
Record Dates: First submitted 2007-03-16; First posted 2007-03-19 (Estimated); Last update posted 2013-07-16 (Estimated); Status verified 2009-04

CONDITIONS: Healthy
Keywords: catechin; oxidative stress; chromosome damage; aged

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (1):
- catechin (Experimental): catechin capsule group
  Interventions: Dietary Supplement: catechin extracts

INTERVENTIONS:
Dietary Supplement: catechin extracts — comparison with placebo

SUMMARY:
The purpose of this study is to clarify the effects of tea catechin extracts on the frequency changes of micronuclei in peripheral lymphocytes compared with other oxidative stress markers in late middle aged healthy volunteers

DETAILED DESCRIPTION:
Experimental studies have revealed that tea catechin extracts induce preventive effects on oxidative stress, but there have been few clinical trials conducted to verify the effects. Also, there have been few clinical markers indicating oxidative damage, and therefore, more accurate and reliable markers have been expected. The study is designed for evaluating the effects of tea catechin extracts on the frequency changes of micronuclei in peripheral lymphocytes as the indicator of oxidative damage, compared with other oxidative stress markers in late middle aged healthy volunteers.

ELIGIBILITY:
Inclusion Criteria:

* aged 40 to 65 years old
* healthy volunteers
* obtained written informed concent before participation

Exclusion Criteria:

* participant who is not able to refrain from drinking tea for 2 weeks during the study
* participant taking supplements or herbal products including folate, vitamin B, C, E, coenzyme Q10, calcium, for 2 weeks before the study
* participant taking supplements or herbal products including folate, vitamin E for 3 months before the study
* participant possessing tea allergy

Ages: 40 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2007-06; Primary Completion 2009-08 (Actual); Study Completion 2012-04 (Actual)

PRIMARY OUTCOMES:
the frequency changes of micronuclei in peripheral lymphocytes | After seven days untervention

SECONDARY OUTCOMES:
the change of markers of oxidative damage, as measured by 8-hydroxyguanosine (8-OHdG), vitamin C, folate, homocysteine | After seven days intervention

CONTACTS AND LOCATIONS:
Overall Officials: Hiroshi Yamada, MD, PhD, Principal Investigator — University of Shizuoka
Locations (1):
- Shizuoka General Hospital, Shizuoka, Shizuoka, Japan